CLINICAL TRIAL: NCT05862324
Title: A Phase 1/2 Study Investigating the Safety and Efficacy of Autologous TAC T Cells in Subjects With Unresectable, Locally Advanced or Metastatic Claudin 18.2+ Solid Tumors
Brief Title: TAC T-cells for the Treatment of Claudin 18.2 Positive Solid Tumors (TACTIC-3)
Acronym: TACTIC-3
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Triumvira Immunologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAC01-CLDN18.2-04
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Solid Tumor
Keywords: Claudin 18.2, Claudin+, Claudin Positive
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: In Phase 1, escalating doses of TAC01-CLDN18.2 will be evaluated to identify the RP2D using the classic 3+3 dose escalation study design. In Phase 2, dose expansion groups will further evaluate the safety, efficacy, and PK of the MTD or RP2D for TAC01-CLDN18.2 in subjects with gastric and esophageal AC (Group A), PDAC (Group B), and ovarian and NSCLC cancers (Group C). In Phase 2, definitions of eligible CLDN18.2+ IHC expression levels will be based on retrospective analysis of data from Phase 1 in association with clinical efficacy because there are no formal CAP/ASCO definitions for CLDN18.2+ IHC expression levels. In Phase 2, a Simon 2-stage design will be used to enroll up to 57 subjects in Group A and 22 subjects in Group C. Group B will enroll up to 10 subjects without a Simon 2-stage design due to its historically low ORRs. The 10 treated subjects in Group B are designed to seek evidence of potential efficacy in this difficult to treat CLDN18.2+ subpopulation of PDAC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAC01-CLDN18.2 (Experimental): Lymphodepletion followed by TAC01-CLDN18.2 as a single IV infusion.
  Interventions: Biological: TAC01-CLDN18.2

INTERVENTIONS:
Biological: TAC01-CLDN18.2 — TAC01-CLDN18.2 preceded by lymphodepletion with fludarabine or clofarabine, cyclophosphamide, and nab-paclitaxel.

SUMMARY:
TAC01-CLDN18.2 is a novel cell therapy that consists of genetically engineered autologous T cells expressing T-cell Antigen Coupler (TAC) that recognizes Claudin 18.2. TAC directs T-cells to the targeted antigen (CLDN 18.2), and once engaged with the target, activates them via the endogenous T cell receptor.

This is an open-label, multicenter Phase ½ study that aims to establish safety, maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D), pharmacokinetic profile and efficacy of TAC01-CLDN18.2.

DETAILED DESCRIPTION:
The TAC technology is a novel approach to modifying T cells, herein referred to as TAC T cells, and using them in the treatment of solid tumors. TAC T cells are produced through genetic engineering, incorporating TAC receptors into a patient's own T cells. This redirects these enhanced T cells to specific cancer antigens, and upon recognition, activates them through the natural signaling pathways of the endogenous TCR.

In the TAC01-CLDN18.2 engineered T cell product; TAC T cells recognize the CLDN18.2, a tight junction protein present on the surface of tumor cells, where the protein expression is no longer limited to tight junctions and are visible to T cells to eradicate them. Consequently, it is hypothesized TAC01-CLDN18.2 will be potentially safe and active in treating patients with CLDN18.2+ solid tumors and provide a clinically meaningful therapeutic benefit in patient populations with high unmet medical need.

This is a first-in-human study investigating TAC01-CLDN18.2 to evaluate the safety, MTD or RP2D, PK, and efficacy in subjects with CLDN18.2+ solid tumors who have been treated with at least 2 lines of prior therapy in Phase 1 and after at least 2 lines and no more than 4 lines of prior therapy in Phase 2 (Note: in each phase, subjects with PDAC may have been treated with 1 line of prior antineoplastic therapy. In addition, subjects who are being treated with current lines of therapy, but not deriving benefit or not tolerating therapy, and have not progressed maybe also eligible as long as they have measurable disease at baseline as a starting reference point). In Phase 1, escalating doses of TAC01-CLDN18.2 will be evaluated to identify the RP2D using the classic 3+3 dose escalation study design.

In Phase 2, dose expansion groups will further evaluate the efficacy, safety, and PK of the MTD or RP2D for TAC01-CLDN18.2 in subjects with gastric and esophageal AC (Group A), PDAC (Group B), and mucinous ovarian and NSCLC cancers (Group C). In Phase 2, definitions of eligible CLDN18.2+ IHC expression levels will be based on analysis of data from Phase 1 for signals of clinical activity since there are no formal CAP/ASCO guidelines for CLDN18.2+ expression levels. In Phase 2, a Simon 2-stage design will be used to enroll up to 57 subjects in Group A and 22 subjects in Group C. Group B (PDAC) will enroll up to 10 subjects as an exploratory cohort due to the historically low ORRs observed in PDAC. The 10 treated subjects in Group B are designed to seek evidence of potential clinical activity in this difficult to treat CLDN18.2+ subpopulation of PDAC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written informed consent obtained before any study procedures are conducted.
2. Age ≥ 18 years at the time of informed consent.
3. Tumor tissue samples positive for CLDN18.2 as assessed by central laboratory.
4. Histologically confirmed advanced, metastatic, unresectable CLDN18.2+ solid tumors after at least 2 lines of prior therapy (Phase 1) and after at least 2 and no more than 4 prior lines of therapy (Phase 2). Subjects with PDAC may have been treated with 1 line of prior therapy.

   1. Subjects with incurable Claudin 18.2 expressing malignancies for which no standard-of-care targeted therapy exists may be enrolled regardless of the number of prior treatment lines.
   2. Specific Phase 1 tumor types include gastric, GEJ, esophageal adenocarcinoma, PDAC, colorectal cancer, cholangiocarcinoma, ovarian mucinous cancer, gallbladder cancer and NSCLC.
   3. Specific Phase 2 tumor types include gastric and esophageal adenocarcinoma (Group A), PDAC (Group B), and ovarian or NSCLC (Group C). Other tumor types are not eligible.
5. Subjects with solid tumors with genetic alterations and mutations (e.g., BRAF, BRCA, EGFR mutations, and ALK translocation) where approved targeted therapies were available to their specific cancers must have been previously treated with such approved therapies, or refused such approved targeted therapy for their cancers, prior to enrollment, or in the opinion of the Investigator would be unlikely to tolerate or derive clinically meaningful benefit from these standard-of-care therapies.
6. Measurable disease per RECIST 1.1 at time of enrollment.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at Screening.
8. Life expectancy of at least 12 weeks.
9. Adequate organ and bone marrow reserve function prior to leukapheresis as outlined in protocol.
10. Recovery to Grade ≤ 1 or baseline for any toxicities due to previous therapy, except alopecia, anemia, thrombocytopenia, neutropenia, and neuropathy.

    1. If a subject received major surgery, they must have recovered from the procedure and/or any complications from the procedure prior to starting TAC01-CLDN18.2 therapy.
    2. Toxicity that has not recovered to Grade ≤ 1 is allowed if it meets the inclusion requirements for laboratory parameters.
11. Adequate vascular access for leukapheresis as per institutional standards
12. For women physiologically capable of becoming pregnant, agreement to use highly effective methods of contraception starting 28 days prior to study treatment and continue for 1 year after the last TAC01-CLDN18.2 infusion. For men who have partners physiologically capable of becoming pregnant, agreement to use an effective barrier contraceptive method and refrain from donating sperm during study treatment and for 1 year after the last TAC01-CLDN18.2 infusion.
13. Subjects who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrollment. Note: Subjects should remain on antiviral therapy throughout study intervention and follow local guidelines for HBV antiviral therapy post completion of study intervention.
14. Subjects with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at Screening. Note: Subjects must have completed curative antiviral therapy at least 4 weeks prior to enrollment.

Exclusion Criteria:

1. Intolerant to any component of TAC01-CLDN18.2
2. Prior treatment with any of the following:

   1. Adoptive cell transfer of any kind, including CAR T cells.
   2. Gene therapy
3. Prior treatment with a CLDN18.2 targeted agent (Phase 2 only)
4. Investigational medicinal product within 5 half-lives or 21 days prior to leukapheresis, whichever is shorter.
5. Participation in or has participated in a study using an investigational device within 4 weeks prior to the first dose of study treatment.
6. Receipt of a live or live-attenuated vaccine within 30 days prior to the first dose of study Intervention. Administration of killed vaccines are allowed.
7. Radiation within 28 days prior to leukapheresis. Palliative radiation is allowed up to 14 days prior to leukapheresis if additional non-irradiated lesions are present.
8. Chemotherapy or targeted small molecule therapy within 14 days prior to leukapheresis, or within 7 days prior to leukapheresis for erlotinib, gefitinib, afatinib, or crizotinib in NSCLC subjects.
9. Colony stimulating factors, including granulocyte-colony stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), erythropoietin, and other hematopoietic cytokines, within 14 days prior to leukapheresis.
10. Immunosuppressive medication within 14 days or corticosteroid treatment < 72 hours prior to leukapheresis, except for physiological replacement doses (< 12 mg/m2/24 hours of hydrocortisone or equivalent) and topical or inhaled steroids.
11. History or presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
12. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study Screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
13. Active inflammatory neurological disorders (e.g., Guillain-Barre Syndrome, amyotrophic lateral sclerosis, multiple sclerosis).
14. Active autoimmune disease (e.g., lupus, rheumatoid arthritis, Sjogren's syndrome) requiring systemic disease modifying agents in the past 2 years. Hormone replacement therapy (e.g., thyroxine, insulin), or physiologic corticosteroid replacement therapy (for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Active or uncontrolled hepatitis B or C (HCV ribonucleic acid [RNA] positive) infection or any history of or active human immunodeficiency virus (HIV) infection.
16. Uncontrolled, acute, or life-threatening bacterial, viral, or fungal infection. Subjects with ongoing use of prophylactic antibiotics, antifungals, or antivirals are eligible if there is no evidence of active infection (includes COVID positive subjects).
17. Class III or IV heart failure (as defined by the New York Heart Association [NYHA]), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease within 6 months prior to Screening.
18. Cardiac arrhythmia not controlled by medical management.
19. Clinically significant thrombotic events within 3 months prior to leukapheresis and/or inability to stop anticoagulation for at least 2 weeks prior to TAC01-CLDN18.2 infusion without compromising a subject's health (except in subjects with PDAC).
20. Prior radiation therapy to the lung > 30 Gy within 6 months of the first dose of study treatment.
21. History of Grade ≥ 3 drug-induced pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
22. Ongoing unstable or active gastrointestinal ulcers and gastrointestinal bleeding.
23. Complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent/recurrent vomiting.
24. History of organ transplantation or awaiting organ transplantation.
25. Known additional malignancy that is progressing or requires active treatment or has been an incurable malignant tumor over the last 5 years. Exceptions include basal cell carcinoma of the skin, non-metastatic squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
26. Pregnancy or lactation. Females physiologically capable of becoming pregnant must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test result at Screening and within 48 hours prior to the first dose of LDC.
27. As determined by the Investigator, any uncontrolled medical, psychological, familial, sociological, or geographical condition(s) that do(es) not permit compliance with the protocol.
28. Has a known psychiatric or any disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 24 Months
  Document incidence of DLTs; Type, frequency, and severity of AEs (including clinically significant laboratory abnormalities).
Phase 2: Evaluate Overall Response Rate (ORR) | 24 Months
  Defined as the percentage of treated subjects with a complete or partial response (CR or PR) as assessed by imaging using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Phase 2: Evaluate Duration of Response (DoR) | 24 Months
  Defined as time from first response to disease progression, end of study, start of another anticancer therapy, or death.
Phase 2: Evaluate Overall survival (OS) | 24 Months
  Defined as time from infusion to death from any cause.
Phase 2: Evaluate Disease control rate (DCR) | 24 Months
  Defined as the percentage of treated subjects with stable disease (SD), PR, and CR as assessed by imaging using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Phase 2: Evaluate Progression-Free survival (PFS) or Time to progression (TTP) | 24 Months
  Defined as time from infusion to disease progression or death from any cause.

SECONDARY OUTCOMES:
Phase 1: Determine MTD or RP2D for TAC01-CLDN 18.2 | Up to 29 Days Post TAC01-CLDN18.2 infusion
  Document incidence of Dose-Limiting Toxicities.
Phase 1: Evaluate Overall Response Rate (ORR) | 24 months
  Defined as the percentage of treated subjects with a complete or partial response (CR or PR) as assessed by imaging using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Phase 1: Evaluate Duration of Response (DoR) | 24 Months
  Defined as time from first response to disease progression, end of study, start of another anticancer therapy, or death.
Phase 1: Evaluate Overall survival (OS) | 24 Months
  Defined as time from infusion to death from any cause. Duration of persistence of TAC T cells
Phase 1: Evaluate Disease control rate (DCR) | 24 Months
  Defined as the percentage of treated subjects with stable disease (SD), PR, and CR as assessed by imaging using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Phase 1: Evaluate Progression-Free survival (PFS) or Time to progression (TTP) | 24 Months
  Defined as time from infusion to disease progression or death from any cause.
Phase 2: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability). | 24 Months
  Document type, frequency, and severity of AEs (including clinically significant laboratory abnormalities).

OTHER OUTCOMES:
Phase 1 and Phase 2: Cmax of TAC01-CLDN18.2 (pharmacokinetics; PK). | 24 Months
  Defined as the maximum concentration of TAC T cells after infusion; assessed by vector copy number.
  Describe profile of soluble immune factors and relationship to cytokine release syndrome (CRS), neurotoxicity, and TAC T cell engraftment
Phase 1 and Phase 2: Tmax of TAC01-CLDN18.2 (PK) | 24 Months
  Defined as the first study day the Cmax is reached; assessed by vector copy number.
Phase 1 and Phase 2: area under the concentration time curve (AUC) of TAC01-CLDN18.2 (PK) | 24 Months
  Calculated using the trapezoid rule; assessed by vector copy number.
Phase 1 and Phase 2: Duration of persistence of TAC T cells (PK) | 24 Months
  Defined as the time between the first measurement of transgene above the limit of detection until the last observed quantifiable level of transgene; assessed by vector copy number.
Phase 1 and Phase 2: Human anti-mouse antibody (HAMA) detection. | 24 Months
  Correlation of HAMA detection with TAC PK and subject response
Phase 1 and Phase 2: Cytokine level detection | 24 Months
  Correlation with adverse events and subject response
Phase 1 and Phase 2: Product manufacturing feasibility/success | Duration of the study
  Number of successful manufacturing of TAC01-CLDN18.2 products per subject leukapheresis samples.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - University of Southern California, Los Angeles, California
  - University of California San Diego, San Diego, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Cancer Center, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No